CLINICAL TRIAL: NCT03931447
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Day Dose Study To Assess The Safety And Tolerability Of JNJ-72537634 In Healthy Participants
Brief Title: A Safety and Tolerability Study of JNJ-72537634 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: CR108615; 72537634IBD1001 (Other: Janssen Research & Development, LLC); 2018-003700-39 (EudraCT Number)
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1: JNJ-72537634 Dose 1 or Placebo (Part 1 - SD) (Experimental): Each participant will receive pretreatment with oral antibiotic; followed by a single day (SD) study intervention of JNJ-72537634 at dose 1 or placebo after overnight fast on Day 1.
  Interventions: Biological: JNJ-72537634; Biological: Placebo
- Cohort 2: JNJ-72537634 Dose 2 or Placebo (Part 1 - SD) (Experimental): Each participant will receive pretreatment with oral antibiotic; followed by a SD study intervention of JNJ-72537634 at dose 2 or placebo after overnight fast on Day 1.
  Interventions: Biological: JNJ-72537634; Biological: Placebo
- Cohort 3: JNJ-72537634 Dose 1 or Placebo (Part 2 - MD) (Experimental): Each participant will receive pretreatment with oral antibiotic; followed by a multiple day (MD) study intervention of JNJ-72537634 at dose 1 or placebo after overnight fast on Day 1 for 14 consecutive days.
  Interventions: Biological: JNJ-72537634; Biological: Placebo
- Cohort 4: JNJ-72537634 Dose 2 or Placebo (Part 2 - MD) (Experimental): Each participant will receive pretreatment with oral antibiotic; followed by a MD study intervention of JNJ-72537634 at dose 2 or placebo after overnight fast on Day 1 for 14 consecutive days.
  Interventions: Biological: JNJ-72537634; Biological: Placebo

INTERVENTIONS:
Biological: JNJ-72537634 — Participants in Cohort 1 and 3 will receive Dose 1 and participants in Cohort 2 and 4 will receive Dose 2 of JNJ-72537634 as oral capsule.
Biological: Placebo — Participants will receive matching placebo as oral capsule in all cohorts.

SUMMARY:
The purpose of the study is to assess the safety and tolerability of JNJ-72537634 compared with placebo in healthy participants after administration of single and multiple day doses.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 30 kilogram per meter square (kg/m^2) (BMI = weight/height^2), inclusive, and a body weight of at least 50 kilogram (kg)
* Be healthy on the basis of physical examination, medical history, vital signs, and 12 lead electrocardiogram (ECG) performed at screening
* Be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant
* Have normal bowel movements, ranging from 1 to 3 times daily to every other day and have normal consistencies according to the Bristol Stool Scale, ranging from 3 to 5 at admission
* All women of childbearing potential must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test on day of admission

Exclusion Criteria:

* History of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, respiratory disease, hepatic or gastrointestinal (GI) disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Has an active systemic or GI acute or chronic infection as determined by appropriate clinical screening and laboratory tests
* If female, has a positive serum pregnancy test at screening, a positive urine pregnancy test at admission, or is lactating prior to study enrollment
* An active cigarette smoker or has quit cigarette smoking within the previous 6 months
* Has a positive urine toxicology screen at screening or at admission for substances of abuse including but not limited to: barbiturates, benzodiazepines, tetrahydrocannabinol (THC), cocaine, opiates, methamphetamines, tricyclic antidepressants (TCA), methadone, 3,4-methylenedioxymethamphetamine (MDMA), oxycodone, and amphetamines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Part 1 Single Day (SD) Dose: Percentage of Participants With Treatment Emergent Adverse Events (TEAE) and Serious Adverse Events (SAE) as a Measure of Safety and Tolerability | Up to 24 Weeks post final dose
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are adverse events (AEs) which will occur up to 24 Weeks that were absent before treatment or that worsened relative to pre-treatment state. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 2 Multiple Day (MD) Dose: Percentage of Participants With TEAE and SAE as a Measure of Safety and Tolerability | Up to 26 Weeks post final dose
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are AEs which will occur up to 26 Weeks that were absent before treatment or that worsened relative to pre-treatment state. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Part 1 SD: Number of Participants With Abnormalities in Vital Signs, Electrocardiogram (ECG) and Clinically Significant Laboratory Findings as a Measure of Safety and Tolerability | Up to 12 Weeks post final dose
  Number of participants with abnormalities in vital signs, ECG and clinically significant laboratory findings will be reported.
Part 2 MD: Number of Participants With Abnormalities in Vital Signs, ECG and Clinically Significant Laboratory Findings as a Measure of Safety and Tolerability | Up to 14 Weeks post final dose
  Number of participants with abnormalities in vital signs, ECG and clinically significant laboratory findings will be reported.

SECONDARY OUTCOMES:
Part 1: Detection and Abundance of JNJ-72537634 | Up to 24 Weeks
  Stool assessment will be done to characterize the presence of JNJ-72537634.
Part 2: Detection and Abundance of JNJ-72537634 | Up to 26 Weeks
  Stool assessment will be done to characterize the presence of JNJ-72537634.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Silber JL, Norman JM, Kanno T, Crossette EM, Szabady R, Menon R, Marko M, Hao LY, Tomsho L, Bhagat S, Yuan A, Olle B, Lamouse-Smith E. A randomized, double-blind, placebo-controlled, single- and multiple-dose phase 1 study of VE202, a defined bacterial consortium for treatment of inflammatory bowel disease: safety and colonization dynamics of a novel live biotherapeutic product in healthy adults. Eur J Gastroenterol Hepatol. 2025 Oct 23. doi: 10.1097/MEG.0000000000003098. Online ahead of print. PMID 41342324